CLINICAL TRIAL: NCT03993171
Title: A Phase 2, Open-Label, Sequential Group, Investigator Blinded Study of Magnetic Resonance Spectroscopy (31P-MRS) to Assess the Effects of CNM-Au8 for the Bioenergetic Improvement of Impaired Neuronal Redox State in Multiple Sclerosis.
Brief Title: 31P-MRS Imaging to Assess the Effects of CNM-Au8 on Impaired Neuronal Redox State in Multiple Sclerosis.
Acronym: REPAIR-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNMAu8.207
Record Dates: First submitted 2019-05-31; First posted 2019-06-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: neurodegeneration; gold; nanoparticle; NAD+; redox; 31P-MRS; multiple sclerosis; magnetic resonance spectroscopy; nanocrystal; NADH; primary progressive multiple sclerosis; relapsing multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: Open Label, Investigator Blinded, Sequential Cohort (max of 2 cohorts amongst the possible 4 interventions)
Masking Description: Research participants and site personnel are not masked to study drug, but will be blinded to study dose for each cohort (single-blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 7.5mg CNM-Au8 (Experimental): 7.5mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: gold nanocrystals
- 15mg CNM-Au8 (Experimental): 15mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: gold nanocrystals
- 30mg CNM-Au8 (Experimental): 30mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: gold nanocrystals
- 60mg CNM-Au8 (Experimental): 60mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: gold nanocrystals

INTERVENTIONS:
Drug: gold nanocrystals — CNM-Au8 is a dark red/purple-colored liquid formulation consisting of a stable suspension of faceted clean surfaced elemental gold nanocrystals in buffered deionized water with a concentration of up to 0.5 mg/mL of gold. The formulation is buffered by sodium bicarbonate present at a concentration of 0.546 mg/mL. There are no other excipients. The drug product is formulated to be taken orally and will be provided in single dose HDPE containers. The study doses vary by the concentration of gold nanocrystals per milliliter in a volume of 60 mL.
  Other Names: CNM-Au8

SUMMARY:
REPAIR-MS is a single-center open label, sequential group, investigator and patient blinded study to assess the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with Multiple Sclerosis (MS) within fifteen (15) years of Screening. The primary endpoint for this study changes from baseline to week 12 in CNS metabolic changes, based on 31P-MRSimaging.

DETAILED DESCRIPTION:
This is a single-center open-label, sequential group, investigator blinded study of the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with relapsing multiple sclerosis (RMS) within fifteen (15) years of Screening. Patients will be screened over up to a 6-week period.Patients who meet inclusion criteria and none of the exclusion criteria may be enrolled into the clinical study. The initial cohort of patients (Cohort 1) will begin treatment at a dose of 15mg or 30mg CNM-Au8. Upon completion of the first Treatment Period, dose(s) will be selected for the subsequent cohort (Cohort 2), based on the results of the 31P-MRS change versus baseline from the first cohort. A total of two treatment cohorts may be studied. Investigators and patients will remain blinded to study dose until the study database is formally locked. All patients will receive daily oral treatment over twelve (12) consecutive weeks during each cohort's Treatment Period.

There will be three study periods per treatment cohort:

1. A (6) six week screening period (Screening Period);
2. A (12) twelve-week treatment period (Treatment Period);
3. A (6) six-week follow-up period (End-of-Study Assessment).

Patients will be contacted by phone to assess safety and tolerability at Week 2. At Weeks 4, 8, and 12 patients will return to the clinic to complete PK, PD, visual acuity testing, and safety assessments. At the Baseline and Week 12 visits patients will complete 31P-MRS, MRI, and OCT imaging assessments, the 9-Hole Peg Test, Timed 25-Foot Walk Test, Visual Acuity (high and low contrast letter/visual acuity) and the Symbol Digit Modalities Test (SDMT). Following treatment discontinuation at Week 12, patients will complete an end-of-study (EOS) visit at Week 18. All patients who are prematurely discontinued from treatment will complete the end-of-study visit 4-weeks after discontinuation.

ELIGIBILITY:
Patients enrolled in Cohort 1 must meet the following Inclusion Criteria:

1. At least 18 years of age and up to 55 years (inclusive) of age at Screening.
2. Clinical diagnosis of Relapsing Multiple Sclerosis (RMS) (meeting McDonald criteria, 2017).
3. Diagnosis of MS no longer than 15 years prior to Screening.
4. Stable treatment with natalizumab, defined as a stable dose maintained at the standard infusion interval of 28-days (±5 days) for at least the prior six (6) months.
5. Stable disease activity based on the Investigator's judgment over the prior three (3) months.
6. Any hematological parameters and/or biochemical parameters that fall outside the Within Normal Limits range at Screening must be assessed as Not Clinically Significant (NCS) and deemed stable or transient in nature.
7. Able to understand and give written informed consent.

Patients enrolled in Cohort 2 must meet the following Inclusion Criteria:

1. Male or female, aged 18 - 70 years or age (inclusive);
2. Diagnosis of primary progressive multiple sclerosis (PPMS) or nonactive secondary progressive multiple sclerosis (SPMS), according to revised 2017 McDonald criteria at the Screening visit;
3. EDSS score at the Screening visit of less than or equal to 6.5 (inclusive);
4. Participants must be taking either B-cell depleting therapy (e.g., ocrelizumab, rituximab) or S1P modulator therapy (e.g., siponimod) with consistent stable dosing for at least 48 weeks prior to the Screening visit;
5. Any hematological parameters and/or biochemical parameters that fall outside the Within Normal Limits range at Screening must be assessed as Not Clinically Significant (NCS) and deemed stable or transient in nature; and
6. Able to understand and give written informed consent.

Patients enrolled in Cohort 1 must meet the following Exclusion Criteria:

1. Patients with a clinical relapse requiring systemic steroid treatment within the prior three (3) months.
2. Patients treated with any other MS therapy other than natalizumab; or treated with clemastine fumarate.
3. Based on the Investigator's judgment, patients with a history of significant other major medical condition that may interfere with the conduct of the study or interpretation of the study results.
4. Based on the Investigator's judgment, patients who may have difficulty complying with the protocol and/or study procedures.
5. History of any clinically significant abnormality in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with study participation.
6. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 109 per liter) or eosinophilia (absolute eosinophil count of

   ≥500 eosinophils per microliter) at Screening.
7. Patients with a prior history of, or positive serological assay for the presence of HIV infection, or laboratory evidence of active or chronic infection with hepatitis C (HCV) or hepatitis B (HBV). Note, participants who have been vaccinated for HBV and have detectable HB antibodies are not excluded unless positive for hepatitis surface antigen (HBsAg).
8. Patients participating in any other investigational drug trial or using an investigational drug (within 12 weeks prior to screening and thereafter).
9. Positive screen for drugs of abuse or known alcohol abuse.
10. Females who are pregnant, have a positive pregnancy test, are nursing, or who plan to get pregnant during the course of this clinical trial or within 6 months of the end of this trial.
11. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control during the study and for 6 months following completion of study participation.
12. Patients with implanted metal objects in their body that may be affected by an MRI procedure.
13. Patients who are claustrophobic or otherwise unlikely to be able to complete the MRI scanning procedures.
14. Patients with a history of gold allergy.
15. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.
16. Any active ophthalmological cause for retinal damage other than MS (e.g. cataracts, uveitis, macular degeneration, macular exudate, macular edema, glaucoma, severe astigmatism, ocular trauma, neuromyelitis optica, ischemic optic neuropathy, congenital nystagmus, retinal detachment, amblyopia, optic disk drusen).
17. Severe refractive defects: refractive errors (-5 dioptres to +5 dioptres or more in either eye or axial eye length >26 mm), hypermetropia (> 5 dioptres; cylinder > 3 dioptres); or based on the Investigator's judgment any other ophthalmic diseases that might confound the study results or optical coherence tomography assessment.
18. PRN use of stimulant medications including: amphetamine, dextroamphetamine, lisdexamfetamine, methylphenidate, or modafinil; however, stimulant medications, taken on a consistent daily dose for at least 12-weeks are allowed. No changes in the dose of any stimulant medications are allowed during the study.

Patients enrolled in Cohort 2 must meet the following Exclusion Criteria:

1. History of MS relapses or gadolinium-enhancing lesions seen on brain MRI scans within the five (5) years prior to the Screening visit.
2. History of AQP4, MOG Ab(+) status, or documented ≥ 3 contiguous segment lesion in the spinal cord.
3. Any diagnosis other than PPMS or SPMS that could explain a participant's signs and symptoms.
4. Participants taking any MS disease-modifying therapy other than Bcell depleting therapy (e.g., ocrelizumab, rituximab) or S1P modulator therapy (e.g., siponimod), or not taking disease modifying therapy.
5. Based on the Investigator's judgment, patients with a history of significant other major medical condition that may interfere with the conduct of the study or interpretation of the study results.
6. Based on the Investigator's judgment, patients who may have difficulty complying with the protocol and/or study procedures.
7. History of any clinically significant abnormality in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with study participation.
8. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥500 eosinophils per microliter) at Screening.
9. Patients with a prior history of, or positive serological assay for the presence of HIV infection, or laboratory evidence of active or chronic infection with hepatitis C (HCV) or hepatitis B (HBV). Note, participants who have been vaccinated for HBV and have detectable HB antibodies are not excluded unless positive for hepatitis surface antigen (HBsAg).
10. Patients participating in any other investigational drug trial or using an investigational drug (within 12 weeks prior to screening and thereafter).
11. Positive screen for drugs of abuse or known alcohol abuse.
12. Females who are pregnant, have a positive pregnancy test, are nursing, or who plan to get pregnant during the course of this clinical trial or within 6 months of the end of this trial.
13. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control during the study and for 6 months following completion of study participation.
14. Patients with implanted metal objects in their body that may be affected by an MRI procedure.
15. Patients who are claustrophobic or otherwise unlikely to be able to complete the MRI scanning procedures.
16. Patients with a history of gold allergy.
17. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
The change from baseline to week 12 in CNS metabolic changes, based on 31P-MRS Redox Ratio. | At 12 Weeks
  Mean change in average NAD+/NADH measured brain Redox Ratio by treatment cohort from Baseline to Week 12.

OTHER OUTCOMES:
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of ATP (a, B, y) by subject per dosing group. | At 12 Weeks
  Mean change in average CNS concentration of ATP (a, B, y) by treatment group.
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of NAD+/NADH pool by subject per dosing group. | At 12 Weeks
  Mean change in average CNS concentration of NAD+/NADH pool by treatment group.
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Phosphocreatine (PCr) by subject per dosing group. | At 12 Weeks
  Mean change in average CNS concentration of pooled Phosphocreatine by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Intracellular inorganic phosphate (Pi(in)) by subject per doing group. | At 12 Weeks
  Mean change in average CNS concentration of intracellular inorganic phosphate by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Extracellular inorganic phosphate (Pi(ex)) by subject per dosing group. | At 12 Weeks
  Mean change in average CNS concentration of extracellular inorganic phosphate by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Uridine Diphosphate Glucose (UDPG) by subject per dosing group. | At 12 Weeks
  Mean change in average CNS concentration of UDPG by treatment group
Mean Change in 31P-MRS Membrane Component Tissue Concentration of Phosphoethanolamine (PE) | At 12 Weeks
  Mean change in average CNS concentration of PE [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Phosphocholine (PC) | At 12 Weeks
  Mean change in average CNS concentration of PC [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of glycerophosphoethanolamine (GPE) | At 12 Weeks
  Mean change in average CNS concentration of GPE [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Glycerophosphocholine (GPC) | At 12 Weeks
  Mean change in average CNS concentration of GPC [mmol/kg] by treatment group
9-Hole Peg Test | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the 9-Hole Peg Test by hand.
Timed 25 foot walk test. | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the Timed 25-Foot Walk Test.
Mean Change in Symbol Digit Modality Test (SDMT) | At 12 Weeks
  Mean change in Symbol Digit Modality Test (SDMT) by treatment group from Baseline to Week 12
EDSS | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the Expanded Disability Status Scale. The scale is rated 0-10 with 0 representing normal neurological function, and 10 representing death.
Mean Change in Optical Coherence Tomography (OCT) Retinal Layers of ganglion cell + inner plexiform layer (GCIPL) | At 12 Weeks
  Mean change in Optical Coherence Tomography (OCT) retinal layers by macular scan of Ganglion Cell + inner plexiform layer (GCIPL).
Mean Change in Optical Coherence Tomography (OCT) Retinal Layer of Outer nuclear layer (ONL). | At 12 Weeks
  Mean change in Optical Coherence Tomography (OCT) retinal layers by macular scan of Outer nuclear layer (ONL).
Mean Change in Optical Coherence Tomography (OCT) Retinal Layer of Inner nuclear layer (INL). | At 12 Weeks
  Mean change in Optical Coherence Tomography (OCT) retinal layers by macular scan of Inner nuclear layer (INL).
Mean Change in Optical Coherence Tomography (OCT) Retinal Nerve Fiber Layer by Peripapillary scan. | At 12 Weeks
  Mean change in Retinal Nerve Fiber Layer by Peripapillary Scan (pRNFL)
Mean Change in Myelin Volume Fraction (MVF) | At 12 Weeks
  Mean change in Myelin volume fraction (MVF) in baseline lesions and in normal appearing white matter (NAWM).
Mean Change in Restricted Volume Fraction (F_R) | At 12 Weeks
  Mean Change in Restricted Volume Fraction (F_R) in baseline lesions and in normal appearing white matter (NAWM).
Mean Change in CSF Volume Fraction (F_CSF) | At 12 Weeks
  Mean change in CSF Volume Fraction (F_CSF) between Baseline and Week 12 MRI
Mean Change in Axonal Volume Fraction (AVF) | At 12 Weeks
  Mean Change in Axonal Volume Fraction (AVF) in baseline lesions and in normal appearing white matter (NAWM).
Mean Change in G-Ratio | At 12 Weeks
  Mean change in g-ratio in baseline lesion and in normal appearing white matter (NAWM) represented as an aggregate measure calculated on a per-voxel basis
Mean Change in G-Ration Susceptibility | At 12 Weeks
  Mean change in the g-ratio susceptibility (ppm) in baseline lesion and in normal appearing white matter (NAWM).
Low contrast letter acuity by eye | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the Low contrast letter acuity (LCLA) by eye.
Clinical Global Impression Scale | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the Clinical global impression scale (CGI).
Patient Global Impression Scale | At 12 weeks
  Mean change from Baseline to Week 12 by treatment cohort for the Patient global impression scale (PGI).
Pharmacokinetic Endpoint | Through 18 weeks
  Samples for the measurement of whole blood concentrations of Au will be collected before (pre-dose) administration of the investigational drug product during the Weeks 4 8, and 12 Visits. PK samples will also be collected during the EOS phase at Weeks 14, 16, and 18.
Pharmacodynamic Endpoint | Through 18 weeks
  Blood and urine samples for the measurement of pharmacodynamic (PD) assays will be collected at Baseline (pre-dose) following the PK collection during the Weeks 4, 8, 12 and the Week 18 EOS visit. An optional CSF collection for PD analysis will occur at the Baseline Visit (pre-dose) and Week 12 for subjects who consent to the procedure. PD samples will be stored for future analyses to be specified in a separate PD Analysis Plan to be completed prior to the study database lock.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sguigna, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No